CLINICAL TRIAL: NCT01200771
Title: Impact of the PET-scan in the Diagnosis Strategy of Fever Unknown Origin or Inflammatory Syndrome in Immunocompetent Patients
Brief Title: Impact of the PET in the Diagnosis Strategy of FUO or Inflammatory Syndrome in Immunocompetent Patients FUO-TEP
Acronym: FUO-TEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I07005 FUO TEP
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Fever
Keywords: FDG-PET/CT; FUO; Chronic Inflammatory syndrome; Fever of unknown origin
MeSH Terms: conditions — Fever; Fever of Unknown Origin | interventions — tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: TEP — Intravenous injection of glucose labeled Fluor 18. The patient remains fasted at least 6 hours before the start of the examination. The review lasted 1 hour, during wich the patient should not move.

SUMMARY:
Fever of unknown origin (FUO) and chronic inflammatory syndrome could be seen in many affections. The diagnostic process is still a challenge and could not be specified yet after several clinical studies performed by trained teams using two levels diagnostic procedures. For this reason, the diagnosis involves many additional and expensive tests such as computed tomography (CT scan), scintigraphic imaging, endoscopy, biopsy. There is no evidence-based recommendation for the diagnostic work-up of FUO or chronic inflammatory syndrome. Positron emission tomography with 2-[18F] fluoro-2-deoxy-D-glucose combined with CT scan (FDG-PET/CT) is widely used in malignant diseases and seems to be promising for the diagnosis of inflammatory disorders. Its role has not been yet clearly defined in the investigation of FUO and chronic inflammatory syndrome.

DETAILED DESCRIPTION:
All patients with FUO and chronic inflammatory syndrome will undergo FDG-PET/CT and conventional morphologic imaging modalities. Results of these two diagnostic procedures in identifying diagnostic clues will be compared.

We assume FDG-PET/CT could be safer and more helpful to reach early final diagnosis in patients with FUO and chronic inflammatory syndrome than conventional morphologic imaging modalities

ELIGIBILITY:
Inclusion Criteria:

* Patient with FUO criteria:

Fever since 3 weeks, Temperature > 38.3°C, No diagnostic after 3 days of hospitalization.

* Patient with periodic fever criteria:

Fever with criteria like FUO, Fever-free intervals, and apparent remission of the underlying disease, At least 3 febrile episodes.

* Inflammatory syndrome without any clinical sign, Important inflammatory syndrome: Erythrocyte sedimentation rate ≥ 50 at the first hour, and elevation of at least one another inflammatory parameter (haptoglobin, orosomucoïd, fibrinogen or C-reactive protein), Evolution since more than 3 weeks, No diagnostic orientation after clinical examination and history-taking, No diagnostic clue after 3 days of hospitalisation.
* Oral informed consent obtained.

Exclusion Criteria:

* Demented patient or unable to receive information on the protocol and to give informed consent.
* Pregnant women, or without contraception.
* Contraindication to iodine examination, gallium scintigraphy or 18FDG TEP-scan.
* Immunodeficient patient.
* Know HIV infection, neutropenic patient and nosocomial fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To assess the contribution of FDG-PET/CT in the early diagnostic work-up of patients with FUO or chronic inflammatory syndrome | 3 month

SECONDARY OUTCOMES:
To establish the role of FGD PET in reaching final diagnosis compared to conventional morphologic imaging modalities including computer tomography and gallium-67 citrate scintigraphy. | 3 months
To evaluate sensitivity and specificity of this diagnostic procedure | 3 months
To analyse the cost effectiveness of this diagnostic approach | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim LY, MD, Principal Investigator — University Hospital, Limoges
Locations (19):
- France (19):
  - Médecine Interne - CHU, Amiens, France
  - Médecine Nucléaire - CHU, Amiens, France
  - Médecine Interne - CHU, Lille, France
  - Médecine Nucléaire et Imagerie Fonctionnelle - CHU, Lille, France
  - Médecine Interne - CHU, Limoges, France
  - Médecine Nucléaire - CHU, Limoges, France
  - Médecine Interne - AP-HP - Hôpital Hôtel Dieu, Paris, France
  - Médecine Nucléaire - AP-HP - Hôpital Hôtel Dieu, Paris, France
  - Médecine Interne - AP-HP - La Pitié Salpétrière, Paris, France
  - Médecine Nucléaire - AP-HP - La Pitié Salpétrière, Paris, France
  - Médecine Interne - AP-HP - Hôpital Cochin, Paris, France
  - Médecine Interne - AP-HP - Hôpital Bichat, Paris, France
  - Médecine Nucléaire - AP-HP - Hôpital Bichat, Paris, France
  - Service des Isotopes - CRLCC Centre Eugène Marquis, Rennes, France
  - Département de Médecine pour adulte - CHU, Rennes, France
  - Médecine Interne - CH, Rodez, France
  - Médecine Nucléaire - CH, Rodez, France
  - Médecine Interne - CHU, Toulouse, France
  - Médecine Nucléaire - CHU, Toulouse, France

REFERENCES:
- [Background] Ly KH, Costedoat-Chalumeau N, Liozon E, Dumonteil S, Ducroix JP, Sailler L, Lidove O, Bienvenu B, Decaux O, Hatron PY, Smail A, Astudillo L, Morel N, Boutemy J, Perlat A, Denes E, Lambert M, Papo T, Cypierre A, Vidal E, Preux PM, Monteil J, Fauchais AL. Diagnostic Value of 18F-FDG PET/CT vs. Chest-Abdomen-Pelvis CT Scan in Management of Patients with Fever of Unknown Origin, Inflammation of Unknown Origin or Episodic Fever of Unknown Origin: A Comparative Multicentre Prospective Study. J Clin Med. 2022 Jan 13;11(2):386. doi: 10.3390/jcm11020386. PMID 35054081